CLINICAL TRIAL: NCT07054541
Title: Clinical Study on Ultrasound-guided Percutaneous Intervention for Atrial Septal Defect With the Assistance of Specialized Instruments
Acronym: NOVA-ASD
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Pan Xiangbin, Principal Investigator, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-2614
Record Dates: First submitted 2025-06-17; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Atrial Septal Defect (ASD)
Keywords: Ultrasound-guided; Percutaneous Intervention; Atrial Septal Defect; Pannawire; PAN Procedure; ASD closure; non fluoroscopic
MeSH Terms: conditions — Heart Septal Defects, Atrial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-guided intervention with assistance of specialized instruments group (Experimental): Patients randomized in this group will undergo percutaneous ASD closure under pure ultrasound guidance in the entire process with assistance of specialized instruments.
  Interventions: Procedure: Ultrasound-guided intervention with assistance of specialized instruments
- fluoroscopy-guided intervention group (Active Comparator): Patients randomized in this group will undergo percutaneous ASD closure under fluoroscopic guidance in the entire process
  Interventions: Procedure: fluoroscopy-guided intervention

INTERVENTIONS:
Procedure: Ultrasound-guided intervention with assistance of specialized instruments — After detailed evaluation, patients randomized in this group will undergo percutaneous ASD closure under pure ultrasound guidance in the entire process with assistance of specialized instruments
  Arms: Ultrasound-guided intervention with assistance of specialized instruments group
Procedure: fluoroscopy-guided intervention — After detailed evaluation, patients randomized in this group will undergo percutaneous ASD closure under fluoroscopic guidance in the entire process
  Arms: fluoroscopy-guided intervention group

SUMMARY:
Atrial septal defect (ASD) is a common congenital heart disease, and percutaneous interventional therapy is the main and effective treatment. Traditional percutaneous closure procedures are performed under fluoroscopic guidance and require contrast agents. A retrospective analysis of over 20,000 adult patients with congenital heart disease revealed that even low-dose radiation exposure was significantly associated with an increased long-term risk of malignancy. Moreover, the use of contrast agents carries the risk of allergic reactions and kidney injury. Radiation and contrast agents not only pose iatrogenic harm to patients but also limit the use of interventional techniques in special populations, such as pregnant women, patients with contrast agent allergies, or those with renal insufficiency.

To achieve radiation-free and contrast-free interventional closure procedures, researchers have developed ultrasound-guided percutaneous interventional techniques, yielding satisfactory treatment outcomes. In some cases, these techniques have even enabled cardiovascular procedures to be performed on an outpatient basis, significantly reducing hospitalization time and costs.

This project proposes a large-sample, multicenter, prospective randomized controlled study to determine whether ultrasound-guided percutaneous intervention for ASD with the assistance of specialized instruments is non-inferior to traditional fluoroscopy-guided procedures, while also offering shorter hospital stays and lower medical expenses.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 2 years
* Diagnosed with secundum-type atrial septal defect (ASD) with a diameter ≥ 6 mm and ≤ 36 mm, accompanied by right heart volume overload
* The distance from the defect margin to the coronary sinus, inferior vena cava, superior vena cava, and pulmonary veins is ≥ 5 mm; the distance to the atrioventricular valve is ≥ 7 mm

Exclusion Criteria:

* Pregnant women
* Contrast agent allergy
* Renal insufficiency
* Associated cardiac malformations requiring surgical intervention
* Right-to-left shunt ASD
* Ostium primum ASD and sinus venosus ASD
* Any severe infection within one month before the procedure
* Intracardiac thrombus

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 666 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Procedural success rate | Immediately after implantation
  Procedural success is defined as completion of the ASD closure without conversion to another guidance method or surgical repair under cardiopulmonary bypass, and with a residual shunt no greater than 2 mm immediately after implantation. Evaluation of the primary endpoint was done by specialized sonographers blinded to the intervention.

SECONDARY OUTCOMES:
Successful closure rate | Immediately after implantation, at 30 days, at 3 months after implantation
  Residual shunt ≤ 2 mm immediately after implantation, at 30 days, at 3 months after implantation
Composite of major adverse events | At 3 months after implantation
  Composite of major adverse events at 3 months, including sudden cardiac death, occluder displacement or dislodgement, pulmonary artery stenosis, descending aortic stenosis, pseudoaneurysm, bleeding requiring blood transfusion, new-onset hypertension, arrhythmia requiring pacemaker implantation or long-term medication, cardiac tamponade, stroke with sequelae.
Composite of minor adverse events | At 3 months after implantation
  Composite of minor adverse events at 3 months, including groin hematoma, transient arrhythmia requiring medication or electrical cardioversion, perioperative allergic reaction, transient ischemic attack (TIA), anemia, postoperative infection.
Procedure time | At discharge (assessed up to 3 months)
  Procedure time is defined as the duration from puncture to withdrawal of the arterial sheath
Days of hospital stay | At discharge (assessed up to 3 months)
  Days of hospital stay
Hospitalization cost | At discharge (assessed up to 3 months)
  Hospitalization cost

CONTACTS AND LOCATIONS:
Overall Officials: Fengwen Zhang, MM, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Chinese Academy of Medical Sciences, Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No